CLINICAL TRIAL: NCT07215013
Title: Acoustic Resonance Therapy for Treatment of Empty Nose Syndrome: A Prospective, Phase 2 Randomized Clinical Trial
Brief Title: Acoustic Resonance Therapy for Treating Empty Nose Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jayakar Nayak, Associate Professor of Otolaryngology - Head & Neck Surgery (OHNS), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JN-ENT-R01
Record Dates: First submitted 2025-10-03; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Empty Nose Syndrome; Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Personalized ART (Experimental): Participants receive personalized ART three times a day for 15 minutes over the study duration.
  Interventions: Device: Personalized ART
- Non-personalized ART (Active Comparator): Participants receive non-personalized ART three times a day for 15 minutes over the study duration.
  Interventions: Device: Non-personalized ART

INTERVENTIONS:
Device: Personalized ART — ART personalized to the patient's exact cranio-facial dimensions. Once dimensions are calculated, ART frequency is calculated by an algorithm that is then transmitted to a headband worn by the patient three times a day.
  Other Names: Sonu
  Arms: Personalized ART
Device: Non-personalized ART — ART frequency randomly transmitted to a headband worn by the patient three times a day.
  Arms: Non-personalized ART

SUMMARY:
This study is to determine whether Acoustic Resonance Therapy (ART), an FDA-approved treatment for standard nasal obstruction, may be helpful in mitigating the debilitating symptoms of Empty Nose Syndrome (ENS), which includes an alternative form of nasal obstruction. ART is a non-invasive treatment that uses sound vibrations to improve nasal congestion and other sinus symptoms. ART works by delivering specific frequencies of sound to the sinonasal cavities (nose and sinuses). These vibrations cause the tissues in the sinuses to resonate, which can help break up mucus and clear blockages, reduce inflammation, and improve airflow.

ELIGIBILITY:
Inclusion Criteria:

* Documented case of Empty Nose Syndrome
* Documented past turbinate reduction surgery

Exclusion Criteria:

* Neurocognitive diagnosis/decline

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2028-07 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change in 6-item ENS-6Q Questionnaire Score | Monthly for up to 2 years
  The ENS6Q refers to the 6-Item Nasal Symptom Questionnaire, which is a tool used to assess nasal symptoms in patients, particularly in the context of conditions like allergic rhinitis, chronic rhinosinusitis, or other nasal disorders. This questionnaire helps clinicians evaluate the severity and impact of nasal symptoms on a patient's quality of life. Each item on the questionnaire is typically rated on a scale (e.g., 0 to 3 or 0 to 4). The total score (range: 0 to 30) is calculated by summing the scores from each item, providing an overall assessment of nasal symptom severity. For both item and total scores, higher scores indicate more severe symptoms. A reduction of 7 points from baseline is considered clinically significant reduction in symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jayakar Nayak, MD, PhD, Principal Investigator — Stanford University; Kai Zhao, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes